CLINICAL TRIAL: NCT04615013
Title: A Phase 1 Study of NBTXR3 Activated by Radiotherapy With Concurrent Chemotherapy for Adenocarcinoma of the Esophagus
Brief Title: NBTXR3, Chemotherapy, and Radiation Therapy for the Treatment of Esophageal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0122; NCI-2020-05329 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0122 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-01; First posted 2020-11-04 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-06

CONDITIONS: Cervical Esophagus Adenocarcinoma; Clinical Stage II Esophageal Adenocarcinoma AJCC v8; Clinical Stage IIA Esophageal Adenocarcinoma AJCC v8; Clinical Stage IIB Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Esophageal Adenocarcinoma AJCC v8; Gastroesophageal Junction Adenocarcinoma; Pathologic Stage II Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage III Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIB Esophageal Adenocarcinoma AJCC v8; Thoracic Esophagus Adenocarcinoma
MeSH Terms: interventions — Capecitabine; Carboplatin; Docetaxel; Fluorouracil; dehydroftorafur; Radiotherapy, Intensity-Modulated; Leucovorin; Oxaliplatin; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (NBTXR3, IMRT, chemotherapy) (Experimental): Patients receive NBTXR3 IT or IN on day 1. Beginning day 15, patients undergo IMRT 5 days per week for 6 weeks for a total of 28 fractions, in the absence of disease progression or unacceptable toxicity. Concurrent with IMRT, patients receive a chemotherapy regimen consisting of either fluorouracil and oxaliplatin with or without leucovorin, oxaliplatin and capecitabine, docetaxel and fluorouracil with or without leucovorin, docetaxel and paclitaxel, or carboplatin and paclitaxel per physician discretion.
  Interventions: Drug: Capecitabine; Drug: Carboplatin; Drug: Docetaxel; Drug: Fluorouracil; Other: Hafnium Oxide-containing Nanoparticles NBTXR3; Radiation: Intensity-Modulated Radiation Therapy; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Capecitabine — Not applicable to this study
  Other Names: Ro 09-1978/000; Xeloda
Drug: Carboplatin — Not applicable to this study
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Docetaxel — Not applicable to this study
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Fluorouracil — Not applicable to this study
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Other: Hafnium Oxide-containing Nanoparticles NBTXR3 — Given IT or IN
  Other Names: NBTXR3
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Drug: Leucovorin — Not applicable to this study
  Other Names: Folinic acid
Drug: Oxaliplatin — Not applicable to this study
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Drug: Paclitaxel — Not applicable to this study
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
The purpose of this Phase I study is to determine the recommended phase 2 dose (RP2D) and safety profile of NBTXR3 activated by radiation therapy with concurrent chemotherapy for the treatment of patients with esophageal adenocarcinoma. NBTXR3 is a drug that when activated by radiation therapy, may cause targeted destruction of cancer cells. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Chemotherapy drugs, such as oxaliplatin, fluorouracil, capecitabine, docetaxel, paclitaxel, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving NBTXR3 activated by radiation therapy with concurrent chemotherapy may help control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the recommended phase II dose (RP2D) of hafnium oxide-containing nanoparticles NBTXR3 (NBTXR3) activated by radiotherapy with concurrent chemotherapy, per standard of care, for treatment naive patients with adenocarcinoma of the esophagus.

SECONDARY OBJECTIVES:

I. To evaluate the safety and feasibility of radiation with NBTXR3 in patients with adenocarcinoma of the esophagus.

II. To evaluate the anti-tumor response of chemoradiation with NBTXR3 in patients with adenocarcinoma of the esophagus.

III. To evaluate time-to-event outcomes after chemoradiation with NBTXR3 in patients with adenocarcinoma of the esophagus.

EXPLORATORY OBJECTIVES:

I. To evaluate the body kinetic profile of intratumorally/intranodally injected NBTXR3.

II. To evaluate time to event outcomes for patients with clinical staging of locally advanced, unresectable disease.

III. To evaluate surgical outcomes in patients who undergo surgery after study treatment.

IV. To evaluate radiomic measurements with outcomes. V. To assess immune-related biomarkers of response.

OUTLINE: This is a dose-escalation study of NBTXR3.

Patients receive NBTXR3 intratumorally (IT) or intranodally (IN) on day 1. Beginning day 15, patients undergo intensity-modulated radiation therapy (IMRT) 5 days per week for 6 weeks for a total of 28 fractions in the absence of disease progression or unacceptable toxicity. Beginning on day 15, concurrent with IMRT, patients receive a chemotherapy regimen consisting of either fluorouracil and oxaliplatin with or without leucovorin, oxaliplatin and capecitabine, docetaxel and fluorouracil with or without leucovorin, docetaxel and paclitaxel, or carboplatin and paclitaxel per physician discretion.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of the cervical or thoracic esophagus or gastroesophageal junction
* Adenocarcinoma of the esophagus stages II-III allowed
* Medically able to receive chemoradiation. Following chemotherapy regimens are allowed:

  * Oxaliplatin and fluorouracil (5-FU) or capecitabine
  * Docetaxel and/or 5-FU or paclitaxel
  * Carboplatin and paclitaxel
* Amenable to undergo the endoscopic ultrasound (EUS) guided injection of NBTXR3 as determined by the investigator or treating physician

  * Patients with lesions for which the EUS scope is not able to traverse the tumor are allowed on this trial as long as an injection can be performed as per treating physician's discretion
* Has at least 1 and up to 4 target lesion(s) in the esophagus that are measurable on cross sectional imaging and repeated measurements (via Response Evaluation Criteria in Solid Tumors [RECIST] version [v] 1.1) at the same anatomical location should be achievable

  * Local nodal disease around the esophagus allowed
  * Nodal target lesions must be >= 15 mm (short axis) based on computed tomography (CT) (slice thickness of 5 mm or less) or magnetic resonance imaging (MRI)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Hemoglobin >= 8.0 g/dL
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine =< 1.5 x upper limit of normal (ULN)
* Calculated (Calc.) creatinine clearance > 30 mL/min
* Glomerular filtration ratio > 40 mL/min per 1.73 m^2
* Total bilirubin =< 2.0 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
* Negative urine or serum pregnancy test =< 7 days of NBTXR3 injection in all female participants of child-bearing potential
* Signed informed consent form (ICF) indicating that participant understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

* Prior radiation or any therapy for the treatment of esophageal cancer
* Prior surgical resection of esophageal tumor
* Esophageal cancer with radiographic evidence of metastases at screening
* At screening, past medical history of:

  * Esophageal fistula
  * Tracheoesophageal fistula
  * Siewert type III tumors
* Evidence of bulky disease and/or abutment of tumor above the carina that may result in tracheoesophageal fistulas as determined by the investigator or treating physician

  * Tumors above the carina without defacement of the fat plane between tumor and the airway are allowed
* Known uncontrolled (grade >= 2) or active esophageal or gastric ulcer disease within 28 days of enrollment
* Known contraindication to iodine-based or gadolinium-based intravenous (IV) contrast
* Active malignancy, in addition to esophageal cancer except for basal cell carcinoma of the skin or non-metastatic low risk prostate cancer definitively treated and relapse free within at least 3 months from time of screening
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, renal failure, cardiac arrhythmia, or psychiatric illness that would limit compliance with treatment
* Known active, uncontrolled (high viral load) human immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection
* Female patients who are pregnant or breastfeeding
* Women of child-bearing potential and their male partners who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period. Acceptable methods of contraception are those that, alone or in combination, result in a failure rate of < 1% per year when used consistently and correctly
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | Up to end of treatment visit (day 85)
  Will be coded and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5 criteria. Descriptive summary tables will be produced, providing the DLTs by initial planned dose level of NBTXR3, initial planned volume of NBTXR3 to be injected, the injected volume, the radiation therapy dose given and the details of the concurrent chemotherapy given.
Maximum tolerated dose and recommended phase 2 dose (RP2D) | Up to end of treatment visit (day 85)
  The Bayesian Optimal Interval design, with accelerated titration, will be used to identify RP2D.

SECONDARY OUTCOMES:
Incidence of NBTXR3/radiation therapy related late onset toxicities | From end of treatment visit (day 85) until end of study (1 year)
  Will be defined as any grade >= 3 adverse event.
Feasibility of NBTXR3 injection in the esophageal tumor and involved regional lymph nodes | Up to 1 year
  The feasibility features of NBTXR3 local administration by intratumoral injection will be presented relative to the initial planned volume level in every cohort.
Objective response rate | Up to 1 year
  Will be defined as the rate of complete or partial response per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, in target and non-target lesions.
Major pathological response rate | Up to 1 year
  Will be assessed by the Modified Ryan Scheme for Tumor Regression Score.
Local progression-free survival | From NBTXR3 injection to locoregional (i.e., within the esophagus or regional nodes) disease recurrence, local progression confirmed radiographically (RECIST v1.1), or death from any cause, whichever occurs first, assessed up to 1 year
  Will be estimated using the method of Kaplan and Meier. Median times and 95% confidence intervals will also be estimated per dose level.
Distant progression-free survival | From NBTXR3 injection to the radiographic confirmation (RECIST version 1.1) of a new lesion outside the esophagus and regional nodes, or death from any cause, whichever occurs first, assessed up to 1 year
  Will be estimated using the method of Kaplan and Meier. Median times and 95% confidence intervals will also be estimated per dose level
Progression-free survival | From NBTXR3 injection to local recurrence, local progression, distant progression, confirmed radiographically (RECIST version 1.1), or death from any cause, whichever occurs first, assessed up to 1 year
  Will be estimated using the method of Kaplan and Meier. Median times and 95% confidence intervals will also be estimated per dose level.
Overall survival | From NBTXR3 injection to death from any cause or end of study, whichever occurs first, assessed up to 1 year
  Will be estimated using the method of Kaplan and Meier. Median times and 95% confidence intervals will also be estimated per dose level.

OTHER OUTCOMES:
Time-course dependent presence of hafnium in blood and urine following NBTXR3 intratumoral/intranodal injection | Up to 4 hrs post NBTXR3 injection
Disease control rate | At 6 months post NBTXR3
  Will be defined as the proportion of patients without progression (local or distant) 6-months post NBTXR3 injection.
R-status | Up to 1 year
  Will be assessed macroscopically by surgeon.
Pathological response rate | Up to 1 year
  Will be assessed by the Modified Ryan Scheme for Tumor Regression Score.
Prognosis of patients with baseline and follow-up quantitative computed tomography image-based analysis | Up to 1 year
Changes in radiomic measurements | Baseline up to 1 year
  Will evaluate clinical and pathological outcomes of patients with changes in radiographic features.
Tumor microenvironment | Up to time of surgery or up to 141 days after end of treatment visit (for patients not undergoing surgery)
  Will analyze the tumor microenvironment through multiplexed immunohistochemistry (mIHC).
Ribonucleic acid expression | Up to time of surgery or up to 141 days after end of treatment visit (for patients not undergoing surgery)
Cytokine profiling | Up to 1 year
Immune activation quantification | Up to 1 year
  Will quantify immune activation by analyzing T and B cells, peripheral blood mononuclear cells using flow cytometry, and esophageal cancer biopsies using mIHC.
Concordance of cell free deoxyribonucleic acid (DNA) | Up to 1 year
  Will evaluate the concordance of cell free DNA detected mutations to those detected in esophageal cancer tumor-derived DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Lin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org